CLINICAL TRIAL: NCT04867655
Title: Acute Effect of Orange Juice Mixed With Oat β-Glucan on Bioavailability of Polyphenols in Healthy Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Dalia Malkova, Senior Lecturer, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Glasgow University
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Healthy
Keywords: Flavanones; β-Glucan; Orange Juice; Biological Availability

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orange juice only (Experimental): Experimental test for 24 hours after consumption of orange juice only (Tropicana 'with bits').
  Interventions: Other: Orange Juice
- Orange Juice mixed with either 6g or 3 g of β-Glucan (Experimental): Experimental test for 24 hours after consumption of orange juice (Tropicana 'with bits') with either 6g or 3 g of β-Glucan.
  Interventions: Other: Orange juice with either 6g or 3 g of β-Glucan

INTERVENTIONS:
Other: Orange Juice — Approximately 500 ml of orange juice will be consumed and then blood and urine samples will be collected for 24 hours
  Arms: Orange juice only
Other: Orange juice with either 6g or 3 g of β-Glucan — Approximately 500 ml of orange juice mixed with either 6g or 3 g of β-Glucan will be consumed and then blood and urine samples will be collected for 24 hours
  Arms: Orange Juice mixed with either 6g or 3 g of β-Glucan

SUMMARY:
Brief summary Orange juice is the most widely consumed fruit juice, accounting for around a third of the total fruit juice market and is a rich source of vitamin C and bioactive compounds, predominantly flavonoids. Current research into the health effects of fruit juice consumption has presented some conflicting conclusions. Although potential health benefits have been attributed to the anti-inflammatory and anti-oxidant properties of the bioactive components in juice, other studies have suggested that the benefits of consuming orange are outweighed by the negative implications of the high sugar content leading to increases in blood glucose and insulin. At the same time it is well established that supplementation with a mean dose of 5g of β-Glucan, a soluble fibre derived from cereals such as oats or barley, significantly reduces insulin and glucose in healthy subjects and metabolic compromised individuals. Thus, the formulation of an OJ beverage with an added β-Glucan supplement may be a useful strategy to attenuate the detrimental impact of high sugar content. However, while delaying the absorption of glucose brings about favourable effects on post-prandial glycemia, dietary fibre may also reduce the bioavailability of some beneficial compounds, including polyphenols. So far, it remains unclear how addition of β-Glucan impacts bioavailability of orange juice flavanones. Thus, this study aims to determine how the bioavailability of orange juice polyphenols of healthy adults is affected mixing orange juice with 3 g and 6 g of oat β-Glucan.

DETAILED DESCRIPTION:
Brief summary Orange juice is the most widely consumed fruit juice, accounting for around a third of the total fruit juice market and is a rich source of vitamin C and bioactive compounds, predominantly flavonoids. Current research into the health effects of fruit juice consumption has presented some conflicting conclusions. Although potential health benefits have been attributed to the anti-inflammatory and anti-oxidant properties of the bioactive components in juice, other studies have suggested that the benefits of consuming orange are outweighed by the negative implications of the high sugar content leading to increases in blood glucose and insulin. At the same time it is well established that supplementation with a mean dose of 5g of β-Glucan, a soluble fibre derived from cereals such as oats or barley, significantly reduces insulin and glucose in healthy subjects and metabolic compromised individuals. Thus, the formulation of an OJ beverage with an added β-Glucan supplement may be a useful strategy to attenuate the detrimental impact of high sugar content. However, while delaying the absorption of glucose brings about favourable effects on post-prandial glycemia, dietary fibre may also reduce the bioavailability of some beneficial compounds, including polyphenols. So far, it remains unclear how addition of β-Glucan impacts bioavailability of orange juice flavanones. Thus, this study aims to determine how the bioavailability of orange juice polyphenols of healthy adults is affected mixing orange juice with 3 g and 6 g of oat β-Glucan.

Eligible participants for this study will be healthy adults aged 18 - 50 years and with a BMI in the normal or overweight to obese range (≥20 kg/m2). Participants will be required to be non-smokers, with a stable weight for the previous 3 months, and not engage in regular strenuous physical activity. Other exclusion criteria will include suffering from any chronic disease, taking any medication, or following a special diet, including being vegetarian and vegan. Before being enrolled in the study, potential participants will attend a health screening session, in which they will complete a health screening and physical activity questionnaire

This study will be a randomised controlled cross-over trial in which each participant will complete two 24-h feeding trials. The experimental trials will be separated by a wash out period of at least 7 days. The order of trials will be randomised for each participant, using a random sequence generator. In the morning of the experimental trial participants will consumed approximately 500ml of OJ (Tropicana 'with bits') without or with Oatwell fibre supplement, providing either 6g or 3 g of β-Glucan. Blood samples and urinary fractions will be collected prior to (baseline) and for 24 hours after consumption of corresponding beverage. Participants will be asked to follow a special polyphenol-free diet and record weighted dietary intake for 2 days preceding each trial and during the day of the experimental trial.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* BMI (20 kg/m2-35 kg/m2)
* non-smoker
* not taking any drug therapies
* normal dietary habits

Exclusion Criteria:

* history of gastrointestinal diseases
* following a special diet
* take vitamin supplements, prebiotics, probiotics
* vegetarian
* engaged in strenuous exercise training
* heavy alcohol consumer
* pregnant or breastfeeding (females)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2022-05-04 (Estimated); Study Completion 2022-05-04 (Estimated)

PRIMARY OUTCOMES:
Plasma pharmacokinetics of naringenin, hesperetin, eriodictyol, isorhamnetin and phenolic acid metabolites including phenylpropionic acids, phenylacetic acid and benzoic acid derivatives | 24 hours
  Change in plasma concentrations collected at base line (0 hours) and 0.5,1, 2, 3,4,5,6,7,8, and 24 hours after ingestion of orange juice
Urinary excretion of naringenin, hesperetin, eriodictyol, isorhamnetin and phenolic acid metabolites including phenylpropionic acids, phenylacetic acid and benzoic acid derivatives | 24 hours
  Change in concentrations in urinary fraction collected at base line (0 hours) and after ingestion of orange juice (0-5, 5-8, 8-10, 10-24 hours)

SECONDARY OUTCOMES:
Body weight | 7 days
  Difference in body weight in kilograms between two experimental trials measured by TANITA scales (TBF-300, Cranela, UK).
Body fatness | 7 days
  Difference in percentage of body fat between two experimental trials measured by TANITA scales (TBF-300, Cranela, UK).
Dietary Intake | 3 days and 24 hours
  Difference in energy/macronutrient intake prior to and during the experimental trails measured from weighted food records

CONTACTS AND LOCATIONS:
Overall Officials: Dale Malkova, PhD, Study Chair — University of Glasgow
Locations (1):
- Human Nutrition, College of Medicine, Veterinary and Life Science, Glasgow, United Kingdom

REFERENCES:
- [Derived] Pereira-Caro G, Almutairi TM, Caceres-Jimenez S, Moreno-Rojas JM, Malkova D, Garcia AL, Crozier A. Bioavailability of orange juice (poly)phenols: beta-glucan-rich oat bran decreases urinary excretion of flavanone phase II metabolites and enhances excretion of microbiota-derived phenolic catabolites. Free Radic Biol Med. 2023 Apr;199:34-43. doi: 10.1016/j.freeradbiomed.2023.02.002. Epub 2023 Feb 9. PMID 36764628